CLINICAL TRIAL: NCT01134926
Title: Phase Study Comparing Between Expectant Management and Misoprostol Treatment for Intra-uterine Residua After Pregnancy Termination, Abortion or Delivery
Brief Title: Non Surgical Management for Uterine Residua After Pregnancy Termination, Abortion or Delivery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The principal investigator left the organization
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0014-10-EMC
Record Dates: First submitted 2010-05-29; First posted 2010-06-02 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Intra-uterine Residua
Keywords: Retained products of conception; residua; misoprostol; expectant management
MeSH Terms: interventions — Misoprostol

ARMS (2):
- intra-uterine residua. expectant management (No Intervention): The patients in this arm will not get any treatment and be followed up by US examinations
- Intra-uterine residua. misoprostol (Experimental): The patients in this arm will be treated with misoprostol at the recruitment day. If there will be sonographic evidence of intra-uterine residua the day after, they'll gat another dose.
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — 8oo mcg intravaginal, second dose after one day if there is no response
  Other Names: cytotec
  Arms: Intra-uterine residua. misoprostol

SUMMARY:
The aim of the study is to find out whether conservative treatment - expectant management or medical therapy using misoprostol is beneficial in the case of uterine residua, and which treatment is better.

DETAILED DESCRIPTION:
Retained products of conception are estimated to occur after approximately 1-6% of pregnancies, probably more often after termination of early pregnancies then after term pregnancy. Complication are abdominal pain, infection, bleeding and for the long term - intrauterine adhesions.Blood clots in the uterine cavity can cause similar complications. The definitive treatment is curettage or hysteroscopy, both of which are carried out under general anesthesia and require an operating theater. Although expectant management and uterotonic drugs are practically used in such situation, they are not described in the literature.This study compare between the outcome of misoprostol treatment and expectant management in the case of intrauterine residua after completion of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women with sonographic examination reveals suspicion of intra-uterine residua after completion of pregnancy
* intrauterine cavity, including endometrium, will be at least 15mm

Exclusion Criteria:

* the need for emergency surgical treatment (curettage)
* fever - at least 38 celsius degree
* women who had medical termination of pregnancy and the examination is after less then 2 weeks since treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
abscence of sonographic finding in the uterine cavity | one week since recruitment
  ofter one week, the patients will undergo an US examination.Failure of management defined as uterine cavity width > 15mm

SECONDARY OUTCOMES:
Complications | Within one week since recruitment
  During the study,there will be collection of data considering pain, bleeding, infection and surgical evacuation.
Woman's satisfaction | One week since recruitment
  At the end of the week, the patient will be asked about her satisfaction with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: yfat kadan, MD, Principal Investigator — haemek medical center
Locations (1):
- HaEmek medical center, Afula, Israel